CLINICAL TRIAL: NCT05692245
Title: Dexamethasone vs Ondansetron as the First-line Antiemetic to Prevent Postoperative Nausea and Vomiting After Cesarean Delivery
Brief Title: Dexamethasone vs Ondansetron After Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Staff, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023P000019
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Nausea and Vomiting, Postoperative; Cesarean Section Complications
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized assignment maintained in a sealed envelop. Study medication provided by a independent party. Investigators remain blinded until completion of analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron (Active Comparator): ondansetron 4 mg intravenous, given once after initiation of anesthesia
  Interventions: Drug: Ondansetron
- Dexamethasone (Active Comparator): dexamethasone 8 mg intravenous, given once after initiation of anesthesia
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Ondansetron — Administered Medication
  Arms: Ondansetron
Drug: Dexamethasone — Administered Medication
  Arms: Dexamethasone

SUMMARY:
The goal of this clinical trial is to compare medications in women having a cesarean delivery. The main question it aims to answer are:

• Which medication is better to use as a first-line prevention agent for nausea and vomiting Participants will rate their nausea, pain and other symptoms after surgery Researchers will compare two drugs, ondansetron and dexamethasone to see if the side effects of pain medications are improved after cesarean.

DETAILED DESCRIPTION:
Cesarean delivery is the most common surgical procedure performed in the United States, with approximately 1.2 million cesarean deliveries performed in 2020.(1) Cesarean delivery is preferentially performed under neuraxial anesthesia (spinal or epidural anesthesia) to allow mothers to be awake during the delivery of their child and to improve maternal safety. Despite the routine use of neuraxial techniques for most cesarean deliveries in the United States, many patients experience nausea and/or vomiting either during surgery (intraoperative nausea and vomiting, IONV) or after surgery (postoperative nausea and vomiting, PONV).

PONV has traditionally been associated with female gender, history of motion sickness, nonsmoking status, and opioid use.(2) Other authors have shown increased PONV risk with younger age, type of surgery, and general anesthesia as opposed to regional or neuraxial anesthesia.(3,4) Intrathecal opioids, are the gold standard for pain relief after cesarean delivery, and are part of the Society for Obstetric Anesthesia and Perinatology's (SOAP) Early Recover After Cesarean (ERAC) guideline. However, these medications have been implicated in increased rates of PONV.(5) Given the prevalence of cesarean delivery and the importance of maternal well-being, prophylaxis of nausea and vomiting remains an important issue to address.

Medications from multiple classes are commonly administered to prevent and treat PONV after cesarean delivery. These include 5-HT3 antagonists, dopaminergic antagonists, corticosteroids, antihistamines, and anticholinergics. Ondansetron, a 5HT3 antagonist, and dexamethasone, a corticosteroid, are among the most commonly administered medications due to their efficacy and long track record of safety during pregnancy. Indeed, the SOAP ERAC guideline recommends that at least two agents from different classes be administered perioperatively to decrease the rates of IONV and PONV.(6) They further suggest metoclopramide for IONV prophylaxis, ondansetron or dexamethasone for PONV prophylaxis.

The safety and efficacy of ondansetron and dexamethasone are further supported by a 2021 Cochrane Systematic review analyzing medical prophylaxis against IONV and PONV in cesarean delivery.(6) Both ondansetron and dexamethasone decreased postoperative nausea (Ond: RR 0.45; 10 RCT, 1340 total subjects; Dex: RR 0.59; 6 studies, 733 women) and vomiting rates (Ond: RR 0.47, 10 studies, 1450 women; Dex: RR 0.68; 7 RCT, 793 women). No adverse events from 5HT3 blocking agents or corticosteroids were identified.

Dexamethasone is intriguing as a first-line agent for cesarean delivery since it may have the added benefit of improved pain control and/or decreased postoperative opioid requirement. Several studies have addressed the role of dexamethasone in pain management. A 2008 study by Jaafarpour et al.(8) found a decrease in composite rates of nausea and vomiting, as well reduction of ~1 point on the VAS pain scale for 24 hours following surgery. Data from other studies have been mixed (9, 10, 11).

In conclusion, there is a gap in knowledge in defining the optimal first-line antiemetic for prophylaxis of PONV in patients undergoing cesarean delivery. The goal of this study is to evaluate the effectiveness of ondansetron vs. dexamethasone on PONV rates and postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women (ASA 2)
* Between 18 and 45 years old
* Singleton term pregnancies
* Scheduled or non-labor cesarean delivery
* Neuraxial (spinal or combined-spinal epidural) anesthesia

Exclusion Criteria:

* Refusal to participate
* Known allergy or contraindication to any medication used in the study
* Significant medical or obstetrical disease (ASA ≥ 3)
* Antiemetic use within 24 hours preceding cesarean delivery
* Insulin dependent diabetes
* Hyperemesis gravidarum or chronic antiemetic use
* History of daily or near-daily steroid use during pregnancy
* Opioid use disorder or other chronic pain syndrome
* Opioid use during pregnancy
* Use of antipruritus medication, pruritic urticarial papules of pregnancy, or cholestasis of pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Severity of Nausea | 24 hours
  Visual analogue score for Nausea scored on a 10 centimeter line

SECONDARY OUTCOMES:
Severity of Vomiting | 24 hours
  Number of times subject vomits
Severity of Pain | 24 hours
  Visual analogue score for Pain scored on a 10 centimeter line

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No